CLINICAL TRIAL: NCT03174054
Title: Evaluation of the Added Value of PSMA-PET Compared With Multi-parametric MRI in the Detection and Classification of Prostate Lesions
Brief Title: The Value of PSMA-PET Compared With Multi-parametric MRI in the Detection Prostate Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, david groshar, Proffesor, Assuta Medical Center
Other Study IDs: 0132-16
Record Dates: First submitted 2017-04-18; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: Men aged 40 and over; multi parametric MRI
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with no clear lesion in PET or MRI: If the clinical suspicion of cancer is low, there will be no biopsy, only follow-up. If the decision is to perform a biopsy on the prostate, it will be performed with transrectal sonar guidance and systematic biopsies will be performed (12 samples will be taken from different areas of the prostate)
- Patients with MRI lesions and overlapping mapping lesions: If MRI and PET are matched, a US FUSION MRI biopsy will be taken between 4-8 samples directly from the lesion as well as other systemic prostate samples according to the surgeon's decision. Will be taken and sent separately to pathology.
  Interventions: Procedure: Biopsy
- Patients with a discrepancy between the PET and MRI: A FUSION approach will be biopsy. Four to eight samples for each lesion, as well as other systemic prostate samples will be taken according to the surgeon's decision, and the samples will be marked and sent separately to the pathology.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsies are part of standard procedures in the patients recruited and will not be done due to this study.
  Groups: Patients with MRI lesions and overlapping mapping lesions; Patients with a discrepancy between the PET and MRI

SUMMARY:
Prostate cancer is a common disease in men. In prostate 35% of biopsies, usually done due to increased PSA levels or clinical suspicion, are false negative, despite malignancy.

Multi-parametric prostate MRI detects malignant neoplasm lesions better than other imaging devices.

A sonar-guided prostate biopsy based on multi-parametric MRI images improves detection of malignancy. Ga68 PSMA-PET test uses a radioactive marker that binds to the prostate's cells and is shown to be a primary prostate tumor site in addition to metastasis.

We believe that the combination of measures from a single Ga68 PSMA and multi-parametric MRI test can lead to further improvement in malignancy, better biopsy guidance, and optimal treatment for the patient.

DETAILED DESCRIPTION:
Prostate cancer is the most common and second leading cause of cancer death in men.

Mostly, patients undergo prostate biopsy whenever abnormal digital rectal examination or elevated prostate specific antigen (PSA) levels have been found. Traditionally, trans-rectal US (TRUS) biopsy is performed using 10-12 needles that are inserted into different areas of the prostate gland. Despite this, up to 35% of prostate cancers are still not diagnosed.

The use of multi-parametric prostate MRI (mnMRI) in which T2-weighted sequence, diffusion weighted imaging (DWI) and dynamic contrast enhanced-imaging (DCE) are used has shown to increase the cancer detection rate of clinically significant lesions and better stratify prostate cancer compared to other modalities(3). A pre-biopsy mnMR can identify suspicious lesions that can be targeted on biopsy. Indeed, the use of MRI- US fusion in which pre-biopsy MR images are incorporated with real time biopsy US images has shown to reduce the number of biopsies performed on patients with low grade cancer and increase the detection of intermediate-high risk subgroups of patients(4).

The introduction of PET/MR with the use of PSMA as a radiotracer offers the potential to add a new biomarker to the well-established mnMRI. Different PSMA metrics such as SUV, metabolic tumor volume (MTV) and kinetic parameters can be correlated with lesion detection rate and Gleason score and help tailoring the precise treatment to patients.

The purpose of the current study is to reveal if PSMA-PET has an added value in the detection and stratification of prostate cancer to the currently used nmMRI.

First Objective: To examine whether PSMA-PET increases detection sensitivity and allows better classification of prostate lesions.

Secondary objective: To check the correlation between PSMA-PET measurements and the various indices of multi-parametrial MRI and the histological results.

The work hypothesis: The PSMA PET MRI measurements will improve the ability to identify and classify prostate lesions and conform to the various MRI measurements Research Methods-

The study population:

Patients who have a clinical suspicion of prostate cancer that will be referred to the prostate multi-parameter MRI before deciding on a prostate biopsy Sampling Method: The study is prospective and will include subjects who meet the criteria for inclusion in a continuous manner. The subjects will undergo a PET MRI PSMA test, followed by a prostate fusion biopsy (up to two weeks after the test) using US fusion technology.

Parameters of the PSMA PET-MR test :

PET Measurements: Quantitative calculation of the absorption of suspicious lesions.

The type of biopsy will depend on the PET MRI results. If a suspicious finding is found according to the PET or MR test or both, the biopsy will be done using the US FUSION MRI, and if a suspicious lesion is not seen, the biopsy will be performed by sonar alone, or not at all.

Sample size: 70 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 40 and over.
2. Patients with clinical suspicion of prostate cancer, referred for multi parametric MRI

Exclusion Criteria:

1. Are unable to perform multi-parameter MRI (eg GFR below 30, metals in the body, claustrophobia, etc.).
2. Can not / want to sign informed consent form.

Ages: 40 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with suspected prostate cancer
Study Population: Men aged 40 and over,with clinical suspicion of prostate cancer, referred for multi parametric MRI .
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
correlation between SUV to PSA levels. | 24 months in relation to each patient baseline
  PET Measurements vs. clinical measurements

CONTACTS AND LOCATIONS:
Overall Officials: David Groshar, MD, Principal Investigator — Head of nuclear medicine unit in Assuta Medical Centers

IPD SHARING:
Plan to Share IPD: No